CLINICAL TRIAL: NCT03053349
Title: Ex Vivo Lung Perfusion in Bergamo Lung Transplant Program: A Prospective Observational Study
Brief Title: Ex Vivo Lung Perfusion in Bergamo Lung Transplant Program
Status: Completed | Type: Observational
Sponsor: Papa Giovanni XXIII Hospital (Other)
Responsible Party: Principal Investigator, Stefania Camagni, MD, Papa Giovanni XXIII Hospital
Other Study IDs: EVLP Bergamo - nr 2016-0194
Record Dates: First submitted 2017-02-09; First posted 2017-02-15 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Ex Vivo Lung Perfusion; Lung Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ex Vivo Lung Perfusion (EVLP) appears to be an effective strategy to expand the lung donor pool by better evaluation and reconditioning of non standard grafts. Today, EVLP is clinical practice at the most active transplant centers in North America and Europe.

The aim of this observational prospective monocentric study is to prove the safety and efficacy of EVLP performed in the setting of Bergamo lung transplant program.

A statistically estimated sample size would not fit with the small numbers of Italian lung transplant activity, so the investigators decided to enrol 10 consecutive recipients of grafts subjected to EVLP.

Non standard grafts from Brain Dead Donors (BDD) and Donors after Cardiac Death (DCD) and standard grafts that will undergo prolonged cold ischemic time will be selected for EVLP.

The donor lung procurement operation will be done in the usual manner. The EVLP procedure will be performed in the operating theater of Papa Giovanni XXIII Hospital. The investigators decided to adopt Toronto protocol since it involves some lung protective strategies. EVLP will proceed over a period of at least 4 and not more than 6 hours.

After 60, 120, 180 and 240 minutes from the start of EVLP the following parameters will be evaluated:

* ratio of the partial pressure of arterial oxygen to fraction of inspired oxygen (PO2/FiO2, mmHg)
* Pulmonary Vascular Resistance (PVR, dine*s/cm5)
* Peak Inspiratory Pressure (PIP, cmH2O) and mean airways Pressure (Pawm, cmH2O)
* dynamic lung Compliance (Cpldyn, ml/ cmH2O)
* ΔPO2 = pulmonary vein PO2 - pulmonary artery PO2 (mmHg). Moreover, after 60 and 240 minutes from the start of EVLP a graft X-ray and a bronchoscopy will be performed.

The lung graft will be accepted for transplantation if, after 240 minutes from the start of EVLP, the following conditions are fulfilled:

* PO2/FiO2 >350 mmHg
* stability or reduction of PVR compared with the measurement at the baseline assessment time point
* stability or reduction of PIP and Pawm compared with the measurement at the baseline assessment time point
* stable or better Cpldyn compared with the measurement at the baseline assessment time point
* ΔPO2 >400 mmHg
* improvement of X-ray imaging compared with that at the baseline assessment time point
* exclusion of oedema and purulent secretions by bronchoscopy. After transplantation the recipients will be followed-up for 1 year according to a scheduled timetable.

Data about the EVLP and transplant procedure and about the characteristics of donors and recipients will be collected in a dedicated electronic Case report form (eCRF) according to Good Clinical Practice.

DETAILED DESCRIPTION:
Ex Vivo Lung Perfusion (EVLP) has been allowing to expand the lung donor pool by better evaluation and reconditioning of non standard grafts. The results of both completed and still recruiting prospective clinical trials show similar short- and long-term post-transplant outcomes with non standard and standard grafts subjected to EVLP and traditionally preserved standard grafts. Today, EVLP is clinical practice at the most active transplant centers in North America and Europe.

The aim of this observational prospective monocentric study is to prove the safety and efficacy of EVLP performed in the setting of Bergamo lung transplant program.

A statistically estimated sample size would not fit with the small numbers of Italian lung transplant activity, so the investigators decided to enrol 10 consecutive recipients of grafts subjected to EVLP.

Non standard grafts from Brain Dead Donors (BDD) and Donors after Cardiac Death (DCD) and standard grafts that will undergo prolonged cold ischemic time will be selected for EVLP. Grafts from donors over the age of 65 and/or with a smocking history of more than 10 pack-year and/or with chronic lung disease and/or with gross gastric aspiration and/or with a diagnosis of established pneumonia will be rejected.

The donor lung procurement operation will be done in the usual manner. After excision, the right and left graft will not be divided and will be packed in ice for transportation.

The EVLP procedure will be performed in the operating theater of Papa Giovanni XXIII Hospital. The investigators decided to adopt Toronto protocol since it involves some lung protective strategies. EVLP will proceed over a period of at least 4 and not more than 6 hours.

After 60, 120, 180 and 240 minutes from the start of EVLP the following parameters will be evaluated:

* PO2/FiO2 (mmHg)
* Pulmonary Vascular Resistance (PVR, dine*s/cm5)
* Peak Inspiratory Pressure (PIP, cmH2O) and mean airways Pressure (Pawm, cmH2O)
* dynamic lung Compliance (Cpldyn, ml/ cmH2O)
* ΔPO2 = pulmonary vein PO2 - pulmonary artery PO2 (mmHg). Moreover, after 60 and 240 minutes from the start of EVLP a graft X-ray and a bronchoscopy will be performed.

The lung graft will be accepted for transplantation if, after 240 minutes from the start of EVLP, the following conditions are fulfilled:

* PO2/FiO2 >350 mmHg
* stability or reduction of PVR compared with the measurement at the baseline assessment time point
* stability or reduction of PIP and Pawm compared with the measurement at the baseline assessment time point
* stable or better Cpldyn compared with the measurement at the baseline assessment time point
* ΔPO2 >400 mmHg
* improvement of X-ray imaging compared with that at the baseline assessment time point
* exclusion of oedema and purulent secretions by bronchoscopy. If the lung graft is considered suitable for transplantation, the EVLP procedure will be stopped as described by Toronto protocol and the right and left graft will be divided and packed for hypothermic preservation until implantation.

After transplantation the recipients will be followed-up for 1 year according to a scheduled timetable.

Data about the EVLP and transplant procedure and about the characteristics of donors and recipients will be collected in a dedicated electronic Case Report Form (eCRF) according to Good Clinical Practice.

ELIGIBILITY:
Recipients' Inclusion Criteria:

* lung transplant candidates who are going to be transplanted with grafts subjected to EVLP
* lung transplant candidates who consent to participate in the study by signing the informed consent form.

Recipients' Exclusion Criteria:

* lung transplant candidates who are going to be transplanted with grafts not subjected to EVLP
* lung transplant candidates who are going to be transplanted with grafts subjected to EVLP but refuse consent for their participation in the study.

Ages: 1 Month to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients on the waiting list for monolateral or bilateral lung transplantation at Bergamo lung transplant center
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2020-12-06 (Actual); Study Completion 2020-12-06 (Actual)

PRIMARY OUTCOMES:
Grade of Primary Graft Dysfunction (PGD) | 72 hours after transplantation
  Classification scheme proposed by the International Society for Heart and Lung Transplantation (ISHLT)

SECONDARY OUTCOMES:
Grade of PGD | 24 and 48 hours after transplantation
  Classification scheme proposed by the ISHLT
Need for ECMO | 1 year after transplantation
  Use of post-operative ECMO to support lung and/or heart function (yes/no)
Length of ICU and hospital stay | 1 year after transplantation
  Length of ICU and hospital stay after transplantation (days)
Duration of mechanical ventilation | 1 year after transplantation
  Duration of mechanical ventilation after transplantation (days)
Incidence of anastomotic airway complications | Up to 12 months after transplantation
  MDS endoscopic standardized grading system for macroscopic central airway complications after lung transplantation
30-day mortality | 30 days after transplantation
  Mortality rate 30 days after transplantation
1-year patient survival | 1 year after transplantation
  Patient survival rate 1 year after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Camagni, MD, Principal Investigator — Papa Giovanni XXIII Hospital; Michele Colledan, MD, Study Director — Papa Giovanni XXIII Hospital
Locations (1):
- Papa Giovanni XXIII Hospital, Bergamo, Italy

IPD SHARING:
Plan to Share IPD: No